CLINICAL TRIAL: NCT03401268
Title: A Pilot Study to Assess Tolerability of Subcutaneous Immunoglobulin Treatment (Hizentra) in Patients Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: Subcutaneous Ig in Allogeneic Stem Cell Transplant Recipients
Acronym: ScIGalloHCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScIG alloHCT
Record Dates: First submitted 2018-01-05; First posted 2018-01-17 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hypogammaglobulinemia
Keywords: hypogammaglobulinemia; allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Agammaglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient cohort (Experimental): The study population will include 24 patients, that are either already on IVIG or are eligible for ScIG as initial Ig replacement, that will undergo Ig replacement with subcutaneous immunoglobulin (ScIG) for a total of 6 months.
  Interventions: Drug: subcutaneous immunoglobulin

INTERVENTIONS:
Drug: subcutaneous immunoglobulin — 24 patients demonstrating hypogammaglobulinemia post allogeneic HCT will be started on ScIG for a total of 6 months. Tolerability of the intervention will be assessed with qualitative questionnaires, as well as a financial analysis regarding the intervention.
  Other Names: ScIG

SUMMARY:
Tolerability of home subcutaneous immunoglobulin (ScIG) for replacement therapy for hypogammaglobulinemia in allogeneic HCT patients. A financial analysis comparing the cost of ScIG with intravenous immunoglobulin (IVIG) will also be performed.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether home subcutaneous immunoglobulin (ScIG) is tolerated as replacement therapy for hypogammaglobulinemia in patients that have undergone allogeneic hematopoietic cell transplantation (alloHCT). Secondary objective is to perform a financial analysis comparing the cost of ScIG with intravenous immunoglobulin (IVIG). The study hypothesis is that home based SCIG treatment is applicable and tolerated well for replacement treatment in alloHCT patients. This will be examined in two sets of patients recruited: A) Patients already on IVIG replacement therapy and B) Newly diagnosed patients with hypogammaglobulinemia. Economic analysis will be performed by comparing the cost with an equal number of patients retrospectively determined to have undergone treatment with IVIG.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients at least 100 days post allogeneic hematopoietic cell transplantation for any benign or malignant hematological disease, from a related or unrelated donor
* Patients who are already established on regular IVIG
* Patients eligible for immunoglobulin replacement with an IgG <7mg/L, or normal IgG total but IgG2 or IgG4 below normal
* Patients with IgG =>7g/L but with at least 2 prior episodes of bacterial infection (proven or suspected eg. sinusitis diagnosed on CT)
* No other medical condition which would preclude treatment with immunoglobulin
* Willing to participate and sign informed consent

Exclusion Criteria:

* Previous serious adverse reaction from IVIG or products from Hizentra (polysorbate)
* Other serious medical or psychiatric disorders which may interfere with the patient's ability to participate in the study, or interfere with study assessment (e.g. advanced congestive heart failure, severe liver disease, renal failure, disease relapse or secondary malignancy, schizophrenia, paranoid psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of home ScIG as replacement therapy for hypogammaglobulinemia in allogeneic transplant patients | 6 months
  Qualitative survey describing tolerability, QOL assessment

SECONDARY OUTCOMES:
Financial analysis of cost of ScIG in allogeneic HCT patients | 1 year
  A cost comparison will be performed between the ScIG population and a retrospectively assessed population of allogeneic HCT patients that received IVIG. This will be assessed by a financial analysis and retrospective chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Fotios V. Michelis, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pasic I, Alanazi W, Dranitsaris G, Lieberman L, Viswabandya A, Kim DDH, Lipton JH, Michelis FV. Subcutaneous immunoglobulin in allogeneic hematopoietic cell transplant patients: A prospective study of feasibility, safety, and healthcare resource use. Hematol Oncol Stem Cell Ther. 2021 Dec;14(4):302-310. doi: 10.1016/j.hemonc.2021.01.001. Epub 2021 Feb 23. PMID 33684377